CLINICAL TRIAL: NCT00550537
Title: A Feasibility Study Investigating Translational Science in Chemotherapy-Naive Patients With Stage IIIb or IV Non-Small Cell Lung Cancer (NSCLC) Treated With the EGFR-TKI, Erlotinib
Brief Title: Proteomic Profiling in Predicting Response in Patients Receiving Erlotinib for Stage IIIB, Stage IV, or Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Leora Horn, MD, Assistant Professor of Medicine, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC-THO-0640; P30CA068485 (NIH); VU-VICC-THO-0640; VU-VICC-070494
Record Dates: First submitted 2007-10-26; First posted 2007-10-30 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer; squamous cell lung cancer; adenosquamous cell lung cancer; bronchoalveolar cell lung cancer; large cell lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma, Bronchiolo-Alveolar; Adenocarcinoma of Lung | interventions — Bevacizumab; Carboplatin; Erlotinib Hydrochloride; Paclitaxel; Gene Expression Profiling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Erlotinib followed by paclitaxel + carboplatin (+ bevacizumab in non-squamous) at the time disease progression.
  Interventions: Drug: bevacizumab; Drug: carboplatin; Drug: erlotinib hydrochloride; Drug: paclitaxel; Genetic: gene expression analysis; Genetic: protein expression analysis; Genetic: proteomic profiling; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: bevacizumab — 15 mg/m2 given through a vein for every 3 weeks
Drug: carboplatin — AUC = 6 given through a vein on day 1 of each cycle.
Drug: erlotinib hydrochloride — 150 mg taken by mouth daily
Drug: paclitaxel — 200 mg/m2 given through a vein on day 1 of each cycle.
Genetic: gene expression analysis — Blood and tissue collection.
Genetic: protein expression analysis — Blood and tissue collection.
Genetic: proteomic profiling — Blood and tissue collection.
Other: laboratory biomarker analysis — Blood and tissue collection.

SUMMARY:
RATIONALE: Studying samples of tumor tissue, blood, and urine in the laboratory from patients receiving erlotinib may help doctors predict how patients will respond to treatment.

PURPOSE: The phase II trial is studying proteomic profiling to see how well it predicts response in patients receiving erlotinib for stage IIIB, stage IV, or recurrent non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To define a pre-treatment tumor proteomic profile that predicts response, stable disease, or progressive disease in patients with stage IIIB, stage IV, or recurrent non-small cell lung cancer treated with erlotinib hydrochloride.

Secondary

* To test and refine a pre-treatment serum proteomic expression pattern that predicts response to erlotinib hydrochloride and/or carboplatin and paclitaxel after failing treatment with erlotinib hydrochloride.
* To test and refine tumor proteomic profiles that predict response to carboplatin and paclitaxel after failing treatment with erlotinib hydrochloride.
* To analyze individual and pattern(s) of erlotinib hydrochloride-induced genomic and proteomic biomarker changes in relation to response or non-response to treatment.
* To correlate the efficacy and toxicity of erlotinib hydrochloride with expression of EGFR, EGFR pathway, ErbB family, and other related biomarkers.
* To determine a set of biomarkers to be evaluated in tumor tissue or surrogate tissues prior to treatment with erlotinib hydrochloride to enable patient selection for therapy.
* To estimate response rate and progression-free and overall survival of patients treated with erlotinib hydrochloride as initial therapy.
* To characterize the safety profile of erlotinib hydrochloride in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral erlotinib hydrochloride once daily until disease progression.

At the time of disease progression, patients receive standard chemotherapy comprising paclitaxel IV over 3 hours and carboplatin IV over 15-30 minutes on day 1. Patients with non-squamous cell non-small cell lung cancer also receive bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for up to 6 courses.

Tumor tissue, plasma, serum, and urine samples are collected at baseline for proteomics analysis.

After the completion of study treatment, patients are followed every 8 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer (NSCLC), meeting 1 of the following criteria:

  * Stage IIIB (with pleural effusion) or stage IV disease
  * Recurrent disease after prior surgery
* Measurable or evaluable disease is desirable but not required
* No untreated symptomatic brain metastases

  * Patients who are neurologically unstable despite radiotherapy for the brain metastases are not eligible
  * No requirement for steroids to control neurological symptoms

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,500/mm³
* Hemoglobin ≥ 9 g/dL
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 2.0 mg/dL
* Total bilirubin ≤ 1.5 mg/dL
* Normal hemostasis by history
* PT/PTT within 0.5 seconds of normal range
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Willing to undergo biopsy procedures
* No known severe hypersensitivity to erlotinib hydrochloride or any of the excipients of this product
* No other concurrent malignancies or malignancies diagnosed within the past 5 years, except basal cell carcinoma or cervical cancer in situ
* No significant cardiac disease, including any of the following:

  * NYHA class III or IV heart disease
  * Uncontrolled dysrhythmia
  * Myocardial infarction within the past 6 months
* No evidence of clinically active interstitial lung disease

  * Chronic stable radiographic changes that are asymptomatic allowed
* No evidence of any other severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
* No evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the trial
* No uncontrolled hypertension

  * Blood pressure must be ≤ 150/90 mmHg on a stable antihypertensive regimen

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 6 months since prior adjuvant chemotherapy
* No unresolved chronic toxicity > CTC grade 2 from prior anticancer therapy (except alopecia)
* More than 30 days since prior non-approved or investigational drugs
* No prior chemotherapy for advanced NSCLC
* No concurrent phenytoin, carbamazepine, rifampin, barbiturates, or St. John's wort
* No concurrent administration of other drugs known to inhibit EGFR
* No other concurrent anti-neoplastic or anti-tumor agents, including chemotherapy, radiotherapy, immunotherapy, or hormonal anticancer therapy
* No other concurrent investigational agents
* Concurrent cardioprotective doses of aspirin, as recommended by the physician, for cardiovascular disease allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2007-10; Primary Completion 2011-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Carbone, M.D., Ph.D., Study Chair — Vanderbilt-Ingram Cancer Center
Locations (7):
- United States (7):
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this trial was October 2007 to July 2011. Participants were recruited at Vanderbilt Medical Center, Emory University, M.D. Anderson Cancer Center, University of Florida - Gainesville.
Pre-assignment Details: 10 participants were consented to participate in this trial, but were determined to be ineligible; 3 participants withdrew from the study prior to beginning treatment; 1 participant progressed before beginning treatment.
Period: Overall Study
Arm/Group | Treatment
Started | 116
Completed | 12
Not Completed | 104
Not completed — Death | 18
Not completed — Adverse Event | 20
Not completed — Disease progression before | 46
Not completed — Withdrawal by Subject | 7
Not completed — Change in treatment plan | 4
Not completed — Other complicating ilness | 3
Not completed — Declining performance status | 2
Not completed — Treated closer to home | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 112
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 102
  More than one race | 1
  Unknown or Not Reported | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 116

OUTCOME MEASURES:

1. Primary Outcome: Pre-treatment Tumor Proteomic Profile as a Predictor of Response, Stable Disease, or Progressive Disease
Time Frame: End of treatment date
Population: Lab data was lost by the collaborating institution, Colorado.
Arm/Group | Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Pre-treatment Serum Proteomic Expression Pattern as a Predictor of Response to Erlotinib Hydrochloride and/or Carboplatin and Paclitaxel After Failing Treatment With Erlotinib Hydrochloride
Time Frame: End of treatment date
Population: Lab data was lost by the collaborating institution, Colorado.
Arm/Group | Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Tumor Proteomic Profiles as Predictors of Response to Carboplatin and Paclitaxel After Failing Treatment With Erlotinib Hydrochloride
Time Frame: End of treatment date
Population: Lab data was lost by the collaborating institution, Colorado.
Arm/Group | Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Analysis of Individual and Pattern(s) of Erlotinib Hydrochloride-induced Genomic and Proteomic Biomarker Changes in Relation to Response or Non-response to Treatment
Description: End of treatment date
Time Frame: End of treatment date
Population: Lab data was lost by the collaborating institution, Colorado.
Arm/Group | Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Correlation of the Efficacy and Toxicity of Erlotinib Hydrochloride With Expression of EGFR, EGFR Pathway, ErbB Family, and Other Related Biomarkers
Time Frame: End of treatment date
Population: Lab data was lost by the collaborating institution, Colorado.
Arm/Group | Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Determination of a Set of Biomarkers to be Evaluated in Tumor Tissue or Surrogate Tissues Prior to Treatment With Erlotinib Hydrochloride to Enable Patient Selection for Therapy
Time Frame: End of treatment date
Population: Lab data was lost by the collaborating institution, Colorado.
Arm/Group | Treatment
Number analyzed (Participants) | 0

7. Secondary Outcome: Response Rate for Erlotinib Initial Therapy in Chemotherapy-naïve Patients With Advanced NSCLC
Description: Number of patients in each response category, per RECIST v1.1, summarized as follows for target lesion criteria (see RECIST v1.1 for additional details): complete response (CR),disappearance of target lesions; partial response (PR), >=30% decrease in sum of longest diameter of target lesions; progressive disease (PD), >=20% increase in sum of LD of target lesions or appearance of new lesions; stable disease (SD), insufficient change in target lesions or new lesions to qualify as either PD or SD. The response rate is calculated as the percentage of PR+CR among patients assessed for response.
Time Frame: Through study completion, an average of 1 year
Population: Total 116 participants, 11 not assessed and 4 not evaluable. 101 assessed for response.
Measure: Mean (95% Confidence Interval); unit: percentage of patients assessed
Groups:
- Patients on Erlotinib Segament: Erlotinib followed by paclitaxel + carboplatin (PC) or paclitaxel + carboplatin + bevacizumab (PC+B) in non-squamous cell at the time disease progression.
  bevacizumab: 15 mg/m2 given through a vein for every 3 weeks
  carboplatin: AUC = 6 given through a vein on day 1 of each cycle.
  erlotinib hydrochloride: 150 mg taken by mouth daily
  paclitaxel: 200 mg/m2 given through a vein on day 1 of each cycle.
  gene expression analysis: Blood and tissue collection.
  protein expression analysis: Blood and tissue collection.
  proteomic profiling: Blood and tissue collection.
  laboratory biomarker analysis: Blood and tissue collection.
Arm/Group | Patients on Erlotinib Segament
Number analyzed (Participants) | 101
percentage of patients assessed | 18.8 [12.4 to 27.5]

8. Secondary Outcome: Progression-free Survival (PFS) for Erlotinib Initial Therapy in Chemotherapy-naïve Patients With Advanced NSCLC
Description: PFS is defined as the time from on erlotinib treatment date to progression or death (whichever comes first) before cross-over to PC or PC+B. For those did not progressed nor died, they were censored at the last follow up (either the off erlotinib treatment date or lost follow up date). The median survival time and 95% confidence interval were estimated using Kaplan-meier method.
Time Frame: Through study completion, an average of 1 year
Population: Total 116 participants. One patient was excluded due to death before erlotinib treatment. Total 115 patients were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Patients on Erlotinib Segament
Number analyzed (Participants) | 115
months | 3.16 [2.70 to 4.57]

9. Secondary Outcome: Number of Patients With Worst-grade Toxicities Per Grade
Description: The intensity of the AE will be graded according to the Common Toxicity Criteria (CTC) of the (US) National Cancer Institute (NCI) - Cancer Therapy Evaluation Program (CTEP) [version 3.0 of December 2003] (Appendix B).
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Time Frame: Through study completion, an average of 1 year
Population: 116 paticipants, one patient was excluded due to death before any treatment. All patients who received erlotinib treatment and experienced an Adverse events.
Measure: Number; unit: participants
Groups:
- Erlotinib Segament: Erlotinib followed by paclitaxel + carboplatin (+ bevacizumab in non-squamous) at the time disease progression.
  bevacizumab: 15 mg/m2 given through a vein for every 3 weeks
  carboplatin: AUC = 6 given through a vein on day 1 of each cycle.
  erlotinib hydrochloride: 150 mg taken by mouth daily
  paclitaxel: 200 mg/m2 given through a vein on day 1 of each cycle.
  gene expression analysis: Blood and tissue collection.
  protein expression analysis: Blood and tissue collection.
  proteomic profiling: Blood and tissue collection.
  laboratory biomarker analysis: Blood and tissue collection.
Arm/Group | Erlotinib Segament
Number analyzed (Participants) | 115
participants
  worst-grade 1 | 18
  worst-grade 2 | 51
  worst-grade 3 | 15
  worst-grade 4 | 1

10. Secondary Outcome: Overall Survival for Erlotinib Initial Therapy in Chemotherapy-naïve Patients With Advanced NSCLC
Description: The overall survival time is defined as the time from on treatment to death. Patients were censored of they were alive at the last follow up date. The median survival time and its confidence interval were estimated using Kaplan-meier method.
Time Frame: Through study completion, an average of 1 year
Population: Total 116 participants. One patient was excluded due to death before any treatment.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Erlotinib Followed by PC; Erlotinib Followed by PC+B; Erlotinib: Erlotinib followed by paclitaxel + carboplatin (PC) or paclitaxel + carboplatin + bevacizumab (PC+B) in non-squamous cell at the time disease progression.
  bevacizumab: 15 mg/m2 given through a vein for every 3 weeks
  carboplatin: AUC = 6 given through a vein on day 1 of each cycle.
  erlotinib hydrochloride: 150 mg taken by mouth daily
  paclitaxel: 200 mg/m2 given through a vein on day 1 of each cycle.
  gene expression analysis: Blood and tissue collection.
  protein expression analysis: Blood and tissue collection.
  proteomic profiling: Blood and tissue collection.
  laboratory biomarker analysis: Blood and tissue collection.
Arm/Group | Erlotinib Followed by PC | Erlotinib Followed by PC+B | Erlotinib
Number analyzed (Participants) | 30 | 27 | 58
months | 12.53 [6.94 to 19.10] | 17.23 [8.19 to 30.20] | 6.08 [3.98 to 12.30]

ADVERSE EVENTS:
Time Frame: Patients were evaluated for adverse events at each study visit for the duration of their participation in the study and for 30 days after the discontinuation of Tarceva. After discontinuation from treatment, patients are followed up for all existing and new AEs for 30 calendar days after the last dose of study drug. All new AEs occurring during that period are recorded and followed to resolution when possible.
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 8/116
Other Adverse Events (participants affected / at risk) | 108/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=116)
Infection (urinary tract) (Infections and infestations) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (pharynx) (Infections and infestations) | 1 (1)
Rash (allergy) (Skin and subcutaneous tissue disorders) | 1 (1)
Infection (port) (Infections and infestations) | 1 (1)
Pulmonary (other) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
iatrogenic pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
worsening pneumothorax and subcutaneous emphysema. (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=116)
Diarrhea (Gastrointestinal disorders) | 59 (96)
Nausea (Gastrointestinal disorders) | 42 (69)
Anorexia (Metabolism and nutrition disorders) | 33 (43)
Constipation (General disorders) | 29 (39)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 25 (26)
Vomiting (Gastrointestinal disorders) | 18 (25)
Mucositis (Gastrointestinal disorders) | 15 (17)
Heartburn (Gastrointestinal disorders) | 13 (16)
Rash (acne/acneiform) (Skin and subcutaneous tissue disorders) | 55 (94)
Rash (desquamation) (Skin and subcutaneous tissue disorders) | 40 (76)
Dry skin (Skin and subcutaneous tissue disorders) | 31 (35)
Alopecia (Skin and subcutaneous tissue disorders) | 30 (35)
Dermatology/Skin (other) (Skin and subcutaneous tissue disorders) | 21 (35)
Itching (Skin and subcutaneous tissue disorders) | 16 (20)
Fatigue (Gastrointestinal disorders) | 60 (105)
Weight loss (Eye disorders) | 22 (23)
Chills (General disorders) | 10 (10)
Joint pain (Musculoskeletal and connective tissue disorders) | 24 (35)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (27)
Limb pain (Musculoskeletal and connective tissue disorders) | 19 (25)
Headache (Nervous system disorders) | 15 (17)
Check pain (Respiratory, thoracic and mediastinal disorders) | 14 (18)
Abdominal pain (Gastrointestinal disorders) | 12 (18)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 35 (54)
Cough (Respiratory, thoracic and mediastinal disorders) | 31 (43)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 12 (14)
Pulmonary (other) (Respiratory, thoracic and mediastinal disorders) | 10 (16)
Hyperglycemia (Metabolism and nutrition disorders) | 31 (59)
Hyponatremia (Metabolism and nutrition disorders) | 27 (51)
Serum glutamic pyruvic transaminase (Metabolism and nutrition disorders) | 23 (41)
Alkaline phosphase (Metabolism and nutrition disorders) | 22 (30)
AST, SGOT (Metabolism and nutrition disorders) | 12 (37)
Bilirubin (Metabolism and nutrition disorders) | 17 (21)
Magnesium, serum low (Metabolism and nutrition disorders) | 14 (22)
Albumin, serum low (Metabolism and nutrition disorders) | 11 (15)
Potassium, serum low (Metabolism and nutrition disorders) | 11 (19)
Sensory alteration (Nervous system disorders) | 25 (38)
Dizziness (Nervous system disorders) | 13 (14)
Mood alteration, depression (Psychiatric disorders) | 12 (15)
Anxiety (Psychiatric disorders) | 9 (9)
Hemoglobin (Blood and lymphatic system disorders) | 34 (59)
Leukocytes (Blood and lymphatic system disorders) | 11 (19)
Platelets (Blood and lymphatic system disorders) | 10 (12)
Visual alteration (Eye disorders) | 11 (14)
Dry eye syndrome (Eye disorders) | 10 (10)
Hemorrhage, nose (Respiratory, thoracic and mediastinal disorders) | 13 (19)
Edema, limb (General disorders) | 16 (19)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 13 (15)
Hypertension (Cardiac disorders) | 11 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes